CLINICAL TRIAL: NCT06482138
Title: Dysfunction of Olfaction After SARS-CoV-2 Infection: Morphological and Histomolecular Investigation of Olfactory Cleft Biopsies and Cytobrushes
Brief Title: Dysfunction of Olfaction After COVID-19 Infection: Morphological and Histomolecular Investigation
Acronym: DysOSMIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University Hospital, Geneva (Other); Max Planck Research Unit for Neurogenetics (Unknown); University Hospital Carl Gustav Carus (Other); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: S67380
Record Dates: First submitted 2024-02-19; First posted 2024-07-01 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Covid19; Olfactory Dysfunction
Keywords: Olfactory Dysfunction; COVID-19; SARS-CoV-2; Anosmia; Hyposmia
MeSH Terms: conditions — COVID-19; Anosmia | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Other): Biopsy and cytobrush during a scheduled structural intervention in general anesthesia
  Interventions: Procedure: Biopsy and Cytobrush
- Olfactory Dysfunction (Other): Biopsy and cytobrush during consultation in local anesthesia
  Interventions: Procedure: Biopsy and Cytobrush

INTERVENTIONS:
Procedure: Biopsy and Cytobrush — Collection of olfactory cleft biopsies and cytobrushes

SUMMARY:
Investigation of the mechanisms of persistent SARS-CoV-2 associated olfactory dysfunction (OD) in patients with well-documented olfactory function. The investigators plan to collect olfactory cleft biopsies and cytobrushes in COVID-19 patients and controls.

DETAILED DESCRIPTION:
An explorative prospective clinical study using human body materials of living post-COVID-19 patients with and without OD, to study the mechanisms of persisting olfactory dysfunction. Patients consult ENT specialist for medical purposes and undergo standard-of-care diagnostics and management. The collected tissues from the olfactory cleft mucosa will be analyzed using single cell RNA sequencing and RNAscope combined with immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* Olfactory Dysfunction group: Presence of evident OD (Parosmia, Threshold-Discrimination-Identification (TDI)-score ≤24, Subjective abnormal quantitative olfactory function; measured by a visual analogue score (VAS) of smell impairment ≥5/10
* Control group: No OD (TDI-score >30.5.)

Exclusion Criteria:

* Presence of concomitant nasal mucosal pathology that might affect olfactory function or bias the study investigations
* Use of anticoagulation therapy
* Allergy to local anesthetics

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of olfactory cleft biopsies | From enrollment of 1 patient until analyzed, 1 month
  Morphological and histomolecular differences between OD and control patients
  * Evaluating tissue pathology:
    * Metaplasia
    * hypertrophy
    * aberrant scar formation
    * apoptosis
    * presence of inflammatory cells [H&E, CD68 and CD3 stainings, RNAscope]
  * Presence of SARS-CoV-2 RNA
  * Percentage of OSNs versus sustentacular cells; maturation of OSNs
Analysis of olfactory cytobrushes | From enrollment of 1 patient until analyzed, 1 month
  Morphological and histomolecular differences between OD and control patients
  * Evaluating tissue pathology:
    * Metaplasia
    * hypertrophy
    * aberrant scar formation
    * apoptosis
    * presence of inflammatory cells [H&E, CD68 and CD3 stainings, RNAscope]
  * Presence of SARS-CoV-2 RNA
  * In the olfactory epithelium: percentage of OSNs versus sustentacular cells; maturation of OSNs

CONTACTS AND LOCATIONS:
Overall Officials: Laura van Gerven, Principal Investigator — UZ/KU Leuven
Locations (7):
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
  - UZ/KU Leuven, Leuven, Vlaams-Brabant
  - AZ Sint-Jan Brugge, Bruges, West-Vlaanderen
- Germany (2):
  - University Hospital Carl Gustav Carus, Dresden, Dresden
  - Max Planck Research Unit for Neurogenetics, Frankfurt am Main, Frankfurt
- Switzerland (2):
  - Hôpitaux Universitaires de Genève, Geneva, Canton of Geneva
  - University of Zurich and University Hospital Zurich, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: No